CLINICAL TRIAL: NCT07310420
Title: Phase 1 Single-arm, Open-label, Multicenter Trial to Evaluate Ovarian Suppression Following Subcutaneous ZOLADEX 10.8 mg in Premenopausal Women With Hormone Receptor Positive (HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Advanced Breast Cancer
Brief Title: A Trial to Evaluate Ovarian Suppression Following Subcutaneous ZOLADEX 10.8 mg in Premenopausal Women With HR+, HER2- Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TerSera Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TER-ZLDX-0101
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Cancer
Keywords: Ovarian Suppression; ZOLADEX; HR+; HER2-; Breast Cancer; Goserelin Implant
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZOLADEX 10.8 mg (Experimental): Participants will receive 10.8 mg ZOLADEX on Day 1 and Day 85.
  Interventions: Drug: ZOLADEX

INTERVENTIONS:
Drug: ZOLADEX — Participants will receive ZOLADEX as a subcutaneous (SC) injection on Day 1 (Week 1), and Day 85 (Week 12) for a total of 2 treatments.
  Other Names: Goserelin implant

SUMMARY:
The primary objective of this trial is to evaluate ovarian suppression following treatment with ZOLADEX 10.8 mg by luteinizing hormone (LH).

DETAILED DESCRIPTION:
The purpose of this study is to assess the degree and consistency of ovarian suppression achieved following administration of ZOLADEX 10.8 mg. Ovarian suppression will be evaluated by measuring LH levels over the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender:

   1. Gonadotropin-releasing Hormone (GnRH) treatment-naïve: Female participants aged 18 to 55 years, inclusive.
   2. GnRH treatment-exposed <6 months: Female participants aged 18 to 55 years, inclusive, if GnRH treatment started within <6 months of signing the informed consent.
2. Advanced or metastatic breast cancer: Histological confirmation of breast cancer with evidence of locally advanced or metastatic disease, which is not amenable to surgical resection or radiation therapy with curative intent per investigator's assessment.
3. HR+: Either estrogen receptor positive (ER+) or progesterone receptor positive (PR+) breast cancer, defined as 1% to 100% of tumor nuclei are positive for ER or PR via immunohistochemistry.
4. HER2-: Via American Society of Clinical Oncology, College of American Pathology (ASCO-CAP) guidelines.
5. Prior treatment:

   1. Participants may have received prior radiotherapy.
   2. Participants may have received or be receiving a cyclin-dependent kinase (CDK) 4/6 inhibitor, a phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha-protein kinase B (PIK3CA-AKT) inhibitor, or bisphosphonates if initiated and at a stable dose for at least 2 weeks before trial enrollment.
   3. GnRH treatment-naïve participants will have no history of GnRH agonist or other endocrine therapy in the advanced/metastatic setting.
   4. GnRH treatment-exposed participants may have received a GnRH agonist or other endocrine therapy provided they had established premenopausal status prior to initiating GnRH agonist therapy, within 6 months prior to trial enrollment.
6. Chemotherapy History:

   a. A participant may have received adjuvant or neoadjuvant chemotherapy in early-stage breast cancer.

   i. Any participant who received prior adjuvant or neoadjuvant chemotherapy are eligible provided the criteria for premenopausal status.

   b. All chemotherapy-related toxicities must have recovered to Common Terminology Criteria for Adverse Events (CTCAE) v6.0 ≤Grade 1 before trial participation, except for alopecia, peripheral neuropathy, or paresthesia (≤Grade 2).
7. Concurrent Medications:

   1. Cyclin-dependent kinase 4/6 (CDK4/6) inhibitors are permitted if initiated and tolerated without ongoing toxicity CTCAE v6.0 >Grade 1 for at least 2 weeks before trial enrollment.
   2. PIK3CA/AKT inhibitors are permitted if started at least 2 weeks before the trial and tolerated without ongoing toxicity CTCAE v6.0 >Grade 1.
   3. Concomitant use of bisphosphonates is permitted if initiated and tolerated without ongoing toxicity CTCAE v6.0 >Grade 1 for at least 2 weeks before trial enrollment.
   4. Concomitant use of endocrine therapy (eg, aromatase inhibitor, fulvestrant, or other FDA-approved selective estrogen receptor degraders [SERDs]) is permitted.
8. Informed consent: Able to understand and willing to provide informed consent and able to comply with the trial procedures and restrictions.
9. Contraceptive use: Female participants may be enrolled if they are:

   1. Practicing true abstinence for at least 28 days prior to investigational product (IP) administration until 30 days after the last IP administration and having a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day -1, OR
   2. Using 2 forms of highly effective nonhormonal contraception, including 1 physical barrier (condom or diaphragm) plus another nonhormonal method (eg, intrauterine device, spermicidals) from Screening or at least 2 weeks prior to IP administration (whichever is earlier) until 30 days after the last IP administration and having a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day -1.
10. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

1. Postmenopausal: Naturally or surgically postmenopausal (regardless of age).
2. Body mass index (BMI): <18 kg/m^2 or >35.0 kg/m^2.
3. Prior surgical or radiation procedures: History of bilateral oophorectomy or prior radiotherapy to the ovaries.
4. Recent radiotherapy:

   1. Radiotherapy for breast cancer within 4 weeks prior to trial enrollment.
   2. All radiotherapy-related toxicities (except alopecia) must have recovered to CTCAE v6.0 ≤Grade 1 before trial enrollment.
5. Radiotherapy during trial: Planned radiotherapy during trial period.
6. Selective estrogen receptor modulator (SERM) use during trial: Participants may not receive tamoxifen or other SERMs during the trial and must discontinue any SERMs prior to enrollment, other endocrine therapies (eg, aromatase inhibitor, fulvestrant, or other FDA-approved SERDs) are allowed.
7. Hypersensitivity: Known hypersensitivity, idiosyncratic, or allergic reactions to goserelin, GnRH, GnRH agonists/analogs, or any trial drug components.
8. Expected survival: Estimated life expectancy <6 months from the start of trial therapy, based on the principal investigator's (PI) clinical judgment.
9. Performance status: ECOG performance status ≥3.
10. Life-threatening disease or metastasis: Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, symptomatic pulmonary lymphangitic spread, symptomatic pleural disease, or any symptomatic brain/leptomeningeal metastases (proven or suspected). Participants with asymptomatic or stable/treated brain metastases are eligible to enroll if neurologically stable and are receiving a stable or decreasing corticosteroid dose at the time of enrollment. Participants with discrete pulmonary parenchymal metastases are eligible if respiratory function is not compromised.
11. Hepatic function:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2×upper limit of normal (ULN) if no liver metastases, or >5×ULN with liver metastases.
    2. Total bilirubin ≥1.5×ULN (≥2.5×ULN for Gilbert's syndrome).
12. Renal function: Creatinine clearance (CrCl) ≤30 mL/min as calculated by the Cockcroft-Gault formula.
13. Hematologic parameters:

    1. Hemoglobin (Hgb) <8.0 g/dL.
    2. White blood cell (WBC) count <3000/mm^3.
    3. Platelets <100,000/mm^3.
14. Other malignancies: Active malignancy within the past 3 years, except for adequately treated basal or squamous cell skin cancer or in situ cervical carcinoma.
15. Concurrent medical conditions: Presence of any severe, uncontrolled, or serious illness, medical condition (including psychiatric/addictive disorders), or clinical finding that could compromise trial adherence, as assessed by the investigator.
16. Investigational drug exposure: Exposure to any investigational drug or device within 30 days prior to trial enrollment.
17. Pregnancy: Participant has childbearing potential with a positive serum pregnancy test or positive urine pregnancy test at Screening or Day 1.
18. Breastfeeding: Participant is currently breastfeeding.
19. Contraceptive use: Sexually active with a male partner and not willing to use nonhormonal contraceptive methods throughout the trial. Exceptions: male partner is vasectomized (provided he is her sole sexual partner, and he has received medical assessment of the surgical success), participant has had bilateral salpingectomy or tubal occlusion hysterectomy.
20. Cardiac conditions:

    1. Corrected QT interval (QTc) using Fridericia's correction (QTcF) >450 ms at Screening.
    2. Uncontrolled or symptomatic heart disease, including:

    i. New York Heart Association (NYHA) Class III or IV heart failure.

    ii. Myocardial infarction within the past 6 months.

    iii. Unstable angina or significant arrhythmias requiring intervention.

    c. Documented congenital QT syndrome.
21. Clinically relevant abnormal medical history or abnormal findings on physical examination, vital signs, echocardiogram (ECG), or laboratory tests at Screening that the investigator judges as likely to interfere with the objectives of the trial or the safety of the participant.
22. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
23. History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within the last 1 year prior to IP administration.
24. Major surgery within 30 days prior to IP dosing or a major surgical procedure planned during the trial.
25. Any other condition that precludes adequate understanding, cooperation, and compliance with trial procedures or any condition that could pose a risk to the participant's safety, as per the investigator's judgment.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with LH Values Below a Specified Threshold at Week 6 | Week 6

SECONDARY OUTCOMES:
Percentage of Participants with LH Values below a Specified Threshold at Weeks 12, 18, and 24 | Weeks 12, 18, and 24
Percentage of Participants with Estradiol (E2) Suppression at Weeks 6, 12, 18, and 24 | Weeks 6, 12, 18, and 24
Percentage of Participants with Absence of Menses at Weeks 6, 12, 18, and 24 | Weeks 6, 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Christine Fredericks, Study Director — TerSera Therapeutics LLC

IPD SHARING:
Plan to Share IPD: No